CLINICAL TRIAL: NCT00728598
Title: Vitreous Levels of Patients With Proliferative Diabetic Retinopathy.
Brief Title: Fractalkine, a CX3C Chemokine, Act as a Mediator of Ocular Angiogenesis
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9561702008
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 2008-08

CONDITIONS: Proliferative Diabetic Retinopathy; Angiogenesis
Keywords: Proliferative diabetic retinopathy; Angiogenesis; Vitreous levels; Vascular endothelial growth factor; Fractalkine; Growth factor

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Vitreous sample and blood sample

GROUPS / COHORTS (3):
- 1: Proliferative diabetic retinopathy, active.
- 2: Proliferative diabetic retinopathy, quiescent.
- 3: Control group. Patients with macular hole or idiopathic epiretinal membrane receiving vitrectomy for their disease.

SUMMARY:
Fractalkine (FKN) is a chemoattractant and adhesion molecule for leukocytes. Angiogenic effect of FKN also has been reported. We investigate FKN-mediated angiogenesis in ocular angiogenic disorders.

DETAILED DESCRIPTION:
Fractalkine (FKN), the sole member of the CX3C chemokine family, is named for its fractal geometry. The CX3C motif, with three amino acids between the two terminal cysteines, makes fractalkine distinct from other chemokines.The structure of fractalkine, a membrane-bound glycoprotein with the chemokines domain atop an extended mucin-like stalk, also is unique.Membrane-bound FKN can be markedly induced on primary endothelial cells by inflammatory cytokines; this form promotes the robust adhesion of monocytes and T lymphocytes. Soluble FKN can be released by proteolysis at an efficient chemotactic activity level for monocytes and T cells. Thus, FKN is a versatile molecule regulating both cell-cell interactions in its membrane-bound form and directed-cell migration in its soluble form. The receptor of FKN, CXC3R1, is a G protein-couple protein, which expresses T lymphocytes, monocytes, natural killer (NK) cells, microglia, and neurons.Sulfation of tyrosine enhances the function of CX3CR1 in cell capture and firm adhesion. Fractalkine is expressed constitutively in the kidney, heart, lung, and brain. Fractalkine has demonstrated an important role in CNS inflammation, cardiac allograft rejection, arteriogenesis, renal disease, psoriasis, and during pregnancy. Silverman et al demonstrated the presence of FKN in normal cultured microvascular endothelial and stromal cells of iris and retina in vitro. Upon inflammatory cytokine stimulation, EC also express FKN and its receptors with FKN secretion in an autocrine manner. In addition to EC chemotaxis and tube formation, FKN is an angiogenic mediator in rheumatoid arthritis. Therefore, we hypothesize that FKN not only participates in ocular inflammatory reactions, but also plays an important role in ocular angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of proliferative diabetic retinopathy.
* who will receive vitrectomy for treatment of disease.

Exclusion Criteria:

* previous ocular surgical history.
* history of uveitis
* history of ocular trauma.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with proliferative diabetic retinopathy, who will receive vitrectomy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 1998-01; Primary Completion 1998-12 (Actual); Study Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Vitreous levels and serum levels of Fractalkine, VEGF, other growth factor. | vitreous sample collected on vitrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Hao Yang, MD, PhD, Principal Investigator — Ophthalmology, National Taiwan University Hospital
Locations (1):
- The department of ophthalmology, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Aiello LP, Avery RL, Arrigg PG, Keyt BA, Jampel HD, Shah ST, Pasquale LR, Thieme H, Iwamoto MA, Park JE, et al. Vascular endothelial growth factor in ocular fluid of patients with diabetic retinopathy and other retinal disorders. N Engl J Med. 1994 Dec 1;331(22):1480-7. doi: 10.1056/NEJM199412013312203. PMID 7526212
- [Background] Petrovic MG, Korosec P, Kosnik M, Hawlina M. Vitreous levels of interleukin-8 in patients with proliferative diabetic retinopathy. Am J Ophthalmol. 2007 Jan;143(1):175-6. doi: 10.1016/j.ajo.2006.07.032. Epub 2006 Sep 1. PMID 17188064